CLINICAL TRIAL: NCT06851936
Title: Developing a Scalable Tobacco Cessation Program for Cancer Survivors and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-CCPS-039; IRB202500401 (Other: University of Florida)
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nicotine Use; Tobacco Use
Keywords: tobacco cessation; AHEC; cancer survivors; tobacco; nicotine
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotine Cessation Program (Experimental)
  Interventions: Behavioral: Nicotine cessation program

INTERVENTIONS:
Behavioral: Nicotine cessation program — All participants will complete a nicotine cessation program designed by Area Health Education Center (AHEC). The focus is on known tobacco cessation techniques and motivations to quit with additional focuses on cancer survivors and caregivers. The program consists of 4 sessions (each session is approximately 60 minutes long) that will be delivered by a Tobacco Treatment Specialist by either videoconference or by telephone. Dyad enrollees (i.e., cancer survivors and their caregiver/family member) will complete sessions together. Participants will also be eligible for free nicotine replacement therapy while on study if medically appropriate.

SUMMARY:
Given the challenges to delivering tobacco cessation treatment in oncology care and the unique challenges faced by individuals attempting to quit tobacco after a cancer diagnosis, scalable cessation programs that are tailored to the experiences of cancer survivors that also integrate caregiver/family support are needed. To address this need, this study will use an intervention that consists of two primary strategies: 1) a tailored cessation program for cancer survivors and family members/caregivers who use tobacco and 2) healthcare provider training.

Healthcare providers will receive training on the AAC model (Ask patients about tobacco use, Advise patients to quit, Connect patients to cessation resources), including materials focused on tobacco cessation in cancer care from the CDC, as well as a brief evidence-based communication skills training based on the C-LEAR (Counsel, Listen, Empathize, Answer, Recommend) approach.

ELIGIBILITY:
Inclusion Criteria:

Cancer Survivors including Current Cancer Patients

* Current self-reported user of any tobacco/nicotine product at time of baseline screening assessment (e.g., cigarettes, e-cigarettes, cigars, dip/chew) in the past month.
* Any history of cancer diagnosis. Subjects currently receiving cancer-related treatments are eligible for enrollment.
* Receiving care from the participating UF Health clinics (Medical Oncology, Urology, and Radiation Oncology).
* Capable of completing study requirements
* Informed consent obtained from the subject and documentation of subject agreement to comply with all study-related processes
* Adults aged ≥18 years

Informal Caregivers/Family Members of Cancer Survivors

* Current self-reported user of any tobacco/nicotine product at time of baseline screening assessment (e.g., cigarettes, e-cigarettes, cigars, dip/chew) in the past month.
* A family member, informal caregiver, or friend of an enrolled cancer survivor receiving care from the participating UF Health clinics as described above
* Capable of completing study requirements
* Informed consent obtained from the subject and documentation of subject agreement to comply with all study-related processes
* Adults aged ≥18 years

Exclusion Criteria:

Cancer Survivors including Current Cancer Patients

* Patients unable to complete the sessions because of language, travel or technology barriers
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Informal Caregivers/Family Members of Cancer Survivors

* Participants unable to complete the sessions because of language, travel or technology barriers
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Program reach for cancer survivors | Baseline
  Determine the reach of the nicotine cessation program used in this study for cancer survivors. This is defined as the proportion of eligible patients enrolled (i.e., agreed to participate and consented) during the study period.

SECONDARY OUTCOMES:
Program reach for caregivers/family members of cancer survivors | Baseline
  Determine the reach of the nicotine cessation program used in this study for caregivers/family members of cancer survivors. This is defined as the proportion of enrolled cancer survivors who also have a family member/caregiver enrolled.
Program effectiveness in tobacco cessation | Either 1 week after nicotine cessation program completion or 8 weeks after baseline assessment for participants who do not complete the program sessions
  Determine the effectiveness of the nicotine cessation program used in this study in tobacco cessation. Tobacco cessation will be measured by self-reported 7-day point prevalence abstinence (i.e., no use of any tobacco product over the previous 7 days).
Program effectiveness in tobacco cessation | Either 3 months after nicotine cessation program completion or 5 months after baseline assessment for participants who do not complete the program sessions
  Determine the effectiveness of the nicotine cessation program used in this study in tobacco cessation. Tobacco cessation will be measured by self-reported 7-day point prevalence abstinence (i.e., no use of any tobacco product over the previous 7 days).
Clinic-level adoption of the study intervention | 18 months
  Determine the clinic-level adoption of the study intervention, which is defined as the proportion of eligible patients enrolled by clinic
Healthcare provider-level adoption of the study intervention | 1-2 weeks
  Determine the healthcare provider-level adoption of the study intervention, which is defined as the proportion of eligible healthcare providers participating in the healthcare provider training for this study.
Participant satisfaction | Either 1 week after nicotine cessation program completion or 8 weeks after baseline assessment for participants who do not complete the program sessions
  Determine participant satisfaction with the nicotine cessation program used in this study, which will be measured using a 4-point Lickert scale.
Participant adherence | 8 weeks after baseline assessment
  Determine participant adherence to the nicotine cessation program used in this study, as measured by the number of sessions completed (out of 4).
Participant perspectives on program feasibility and acceptability | Up to 4 weeks after program completion
  Assess participant perspectives on program feasibility and acceptability, using qualitative interviews.
Healthcare provider perspectives on intervention feasibility and acceptability | 18 months
  Assess healthcare provider perspectives on intervention feasibility and acceptability, using qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer LeLaurin, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States